CLINICAL TRIAL: NCT01538316
Title: Clinical Trial on the Effectiveness of the Flavonoids Genistein and Quercetin in Men With Rising Prostate-specific Antigen
Brief Title: Prostate Cancer Prevention Trial With Quercetin and Genistein
Acronym: QUERGEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hohenheim (Other)
Collaborators: University Hospital Tuebingen (Other); Quercegen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, MD, Professor of Medicine, University of Hohenheim
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: ZEM 21 AII
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Primary Prevention of Prostate Cancer
Keywords: Prostate cancer; dietary supplements; quercetin; genistein; prostate-specific antigen; oxidative Status
MeSH Terms: conditions — Prostatic Neoplasms | interventions — genistein combined polysaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Quercetin supplement (Active Comparator)
  Interventions: Dietary Supplement: Quercetin supplement
- Genistein supplement (Active Comparator)
  Interventions: Dietary Supplement: Genistein supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin supplement — 500 mg/d quercetin (+ vitamin C + folic acid + vitamin B3) over a period of six months; crossover design (6 month-periods): followed by genistein and placebo supplement.
  Other Names: Q-Force Chew
  Arms: Quercetin supplement
Dietary Supplement: Genistein supplement — 100 mg/d genistein (+ vitamin C + folic acid + vitamin B3) over a period of six months; crossover design (6 month-periods): followed by placebo and quercetin supplement.
  Other Names: Q-Force Chew
  Arms: Genistein supplement
Dietary Supplement: Placebo — vitamin C + folic acid + vitamin B3 over a period of six months; crossover design (6 month-periods): followed by quercetin and genistein supplement.
  Other Names: Q-Force Chew
  Arms: Placebo

SUMMARY:
The aim of the randomized controlled double-blind crossover trial is to evaluate the effectiveness of two dietary supplements containing polyphenolic phytochemicals (isoflavonoid genistein and flavonoid quercetin) in comparison with placebo on the rate of increase in prostate-specific antigen (PSA). In addition, secondary objective is to evaluate the incidence of prostate cancer and to analyze malondialdehyde and protein carbonyle as indicators of the oxidative status.

DETAILED DESCRIPTION:
Prostate cancer (PC) is the most frequently occurring cancer in men. Its clinical incidence and mortality rates vary geographically, being much lower in Asia than in Western countries. Notably, latent PCs seem to be equally distributed, thus supporting the hypothesis, that environmental factors may be important in prostate cancer progression. Moreover, epidemiological evidence strongly supports the concept that the incidence of clinical prostate cancer depends on lifestyle factors, mainly related to diet. The isoflavone genistein and the flavonoid quercetin have been identified as likely preventive candidates. The aim of the intended clinical trial is to evaluate the hypothesized effectiveness of polyphenolic phytochemicals with highly purified dietary supplements in patients at high risk of clinical PC and without systemic treatment. This will provide data, which serve as an important pre-requesite for targeted dietary interventions using alternative medicine as preventive measures in men with latent PC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with deviant PSA constellation:

  1. Patients with PSA 2,5 - 4 μg/l and free PSA/total PSA < 15 %
  2. Patients with PSA > 4 μg/l with negative punch biopsy of the prostate

     Exclusion Criteria:
* chronic liver diseases, impaired kidney function
* inflammatory diseases of the urogenital tract
* history of malignancy of any organ system, treated or untreated, within the past three years whether or not there is evidence of local recurrence or metastases
* therapy with Doxazosin, Dutaserid and/ or Finasterid, Testosteron and other hormonal active medicaments
* inflammatory bowel diseases
* malabsorption/-digestion
* hypersensitivity/allergy to soy
* phytotherapy or intake of dietary supplements
* smoker
* abnormal clinical laboratory values at baseline
* participation in any other trial with an investigational new drug
* inability to sign informed consent

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Increase in prostate-specific antigen | Every three months (over a period of 18 months)
  Effect on the slope of the regression line though all log2-transformed PSA measurements during the concerned period

SECONDARY OUTCOMES:
Prostate cancer incidence | over the whole study period of 18 months
Quercetin- and genistein blood concentrations | Every three months (over a period of 18 months)
IPSS (International Prostate Symptom Score) | Every three months (over a period of 18 months)
Quality of Life | Every three months (over a period of 18 months)
  SF 36

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, MD, Prof., Study Director — University of Hohenheim; Arnulf Stenzl, MD, Prof., Study Director — Dept. of Urology, University Hospital Tübingen, Germany
Locations (2):
- Germany (2):
  - Institute of Nutritional Medicine, University of Hohenheim, Stuttgart
  - Department of Urology, University Hospital Tübingen, Tübingen